CLINICAL TRIAL: NCT07217977
Title: An Investigational Study Examining the Efficacy of QbMobile in Treatment Monitoring in Individuals With ADHD
Status: Enrolling by invitation | Type: Observational
Sponsor: Qbtech AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 00082513/QB24-02
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD); Attention Deficit Disorder (ADD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
The current study will investigate if QbMobile can be used to improve the accuracy and objective identification of reduced ADHD symptoms in tests scores once treatment has been initiated.

DETAILED DESCRIPTION:
This 4-week study will evaluate QbMobile's performance in monitoring ADHD treatment response. Participants will complete the 10-minute QbMobile test on their personal device during a scheduled clinical visit. They will then repeat the test remotely the following day before beginning their ADHD medication treatment. At week 2 and week 4, participants will take QbMobile remotely at least 1 hour after taking their ADHD medication and no longer than 4 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent (including parent/legal guardians consent when this is required for individuals under 18 years old and assent as is required based on the age of participant) for QbMobile;
* Aged > 6 years and < 60 years old;
* Referred for an ADHD assessment or has a diagnosis of ADHD but not currently receiving any type of stimulant or nonstimulant medication treatment;
* Meets DSM-5 or ICD-11 criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactivity/impulsive presentation) per sites standard clinical care evaluation;
* Qbtech Rating Scale total score of >24 at Visit 1;
* Have adequate sensory and physical ability to complete QbMobile;
* Possess or has access to an iPhone model that supports QbMobile.

Exclusion Criteria:

* Intellectual disability designated by IQ<75);
* Has used psychostimulant medication within 7 days prior to Visit 1;
* A concurrent medical diagnosis that could significantly affect test performance (brain injuries, Parkinson's disease, current epilepsy or active seizures, amyotrophic lateral sclerosis (ALS), multiple sclerosis, dementias (e.g., vascular dementia, Alzheimer disease, etc);
* Other conditions that could affect test performance (migraine or other types of severe headache, chronic or acute pain);
* Substance use (e.g., alcohol, drugs) that may affect performance on the day of the test.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be selected from referrals or participating site's ADHD data base.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in QbMobile Total Score from Baseline at Visit 3 and Visit 4 | Baseline, Visit 3 (Week 2), and Visit 4 (Week 4)
  Change in the QbMobile Total Score from baseline (Visit 2) will be assessed at Visit 3 and Visit 4 to evaluate treatment related responses over time. The QbMobile produces a Total Score number ranging from 0 to 100, where 0 indicates a low likelihood of exhibiting ADHD symptoms and 100 indicates a high likelihood of exhibiting ADHD symptoms. This score is automatically generated in a standard report immediately upon completion of QbMobile.

SECONDARY OUTCOMES:
Change in QbMobile SD-scores from Baseline at Visit 3 and Visit 4 | Baseline, Visit 3 (Week 2), and Visit 4 (Week 4)
  Change in the QbMobile SD-scores (Standard Deviation scores) from baseline (Visit 2) will be assessed at Visit 3 and Visit 4 to evaluate treatment-related effects over time. QbMobile SD-scores are standardized metrics derived from the main parameters (attention, impulsivity, activity and movement). These scores are calculated using and age and sex at birth adjusted normative dataset. The SD-scores are produced in the QbMobile report generated after completion of QbMobile.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Focus-MD, Mobile, Alabama
  - Prodigy Psychiatric Group, San Jose, California
  - Bokhari Medical Consortium, Largo, Florida
  - Nona Pediatric Center, Orlando, Florida
  - Godwin Psychiatry, Goldsboro, North Carolina
  - MindWell Urgent Care, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the research, limited access to supporting data may be granted upon reasonable request under confidentiality agreements from the corresponding sponsor.